CLINICAL TRIAL: NCT02926183
Title: Phase II Study of Neoadjuvant Chemotherapy of Gemcitabine+Nab-paclitaxel Therapy for Patients With Borderline Resectable Pancreatic Cancer
Brief Title: Study of NAC of GA Therapy for Patients With BRPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, NAC-GA investigator, Wakayama Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1881
Record Dates: First submitted 2016-09-27; First posted 2016-10-06 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine plus nab-paclitaxel (Experimental): Neoadjuvant chemotherapy of gemcitabine plus nab-paclitaxel: Enrolled patients were administered a 30-min intravenous infusion of nab-paclitaxel at a dose of 125 mg/m2, followed by a 30-min intravenous infusion of gemcitabine at a dose of 1000 mg/m2, on day 1, 8, and 15 evey 4 weeks as one cycle of regimen.
  Interventions: Drug: Neoadjuvant chemotherapy of gemcitabine plus nab-paclitaxel

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy of gemcitabine plus nab-paclitaxel — Enrolled patients were administered a 30-min intravenous infusion of nab-paclitaxel at a dose of 125 mg/m2, followed by a 30-min intravenous infusion of gemcitabine at a dose of 1000 mg/m2, on day 1, 8, and 15 evey 4 weeks as one cycle of regimen.
  Other Names: NAC-GA for BRPC

SUMMARY:
Gemcitabine plus nub-paclitaxel (GA) regimen was recently presented at an international oncology meeting and represents a new standard regimen in the treatment of metastatic pancreatic cancer. Therefore, it was decided to consider the balance of safety and efficacy on survival time as a preoperative chemotherapy, the investigators use the NAC-GA regimen includes only two cycles (three times weekly and one week rest) of GA regimen.

DETAILED DESCRIPTION:
Gemcitabine plus nub-paclitaxel (GA) regimen was recently presented at an international oncology meeting and represents a new standard regimen in the treatment of metastatic pancreatic cancer. GA is one of the high response rate treatment regimen, the investigators considered as a promising treatment as neoadjuvant chemotherapy. On the other hand, incidences of grade 3 or 4 neutropenia, febrile neutropenia and peripheral neuropathy were significantly higher in the g group compared with gemcitabine group. Therefore, it was decided to consider the balance of safety and efficacy on survival time as a preoperative chemotherapy, the investigators use the NAC-GA regimen includes only two cycles (three times weekly and one week rest) of GEMABR regimen. The investigators also evaluate Recurrence free survival from the first day of protocol therapy, safety of the protocol therapy(Adverse effect), morbidity based on Clavien Dindo classification of more than Grade 3, response rate, preoperative/postoperative tumor marker (CA19-9, CEA), rate of mornalization, reduction rate of SUVmax value on PET-CT (limited only for PET-CT available institutions), chemotherapeutic effect grade based on Evans classification, resection rate, R0 resection rate, surgical data (operative time, blood loss, transfusion, postoperative hospital day), the overall morbidity rates (Reoperation, rate of re-admission, mortality), number of patient rate in postoperative adjuvant therapy (entry rate, completion rate), dose intensity for borderline resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically diagnosed as pancreatic adenocarcinoma, and consistent with NCCN guideline (Version 2. 2016) borderline resectable-arterial, borderline resectable-venous
2. Case with measurable lesion
3. First line treatment
4. PS (ECOG) 0-1
5. >= 20 years old and <80 years old
6. The following criteria must be satisfied in laboratory tests within 14 days of registration

   * WBC count<=12,000/mm3
   * Neutrophil count>=1,500/mm3
   * Hb >= 9.0g/dl
   * Plt >= 100,000/mm3
   * T.Bil <2.0mg/dl (<3=.0mg/dl in biliary drainage case)
   * Serum Cr<=upper limits of normal (ULN)
   * AST, ALT <= 2.5xULN
7. Written informed consent to participate in this study

Exclusion Criteria:

1. Severe drug hypersensitivity
2. Multiple primary cancers within 5 years
3. Severe infection
4. With grade2 or more severe peripheral neuropathy
5. Interstitial pneumonia or pulmonary fibrosis
6. With uncontrollable pleural effusion or ascites
7. With uncontrollable diabetes mellitus
8. With uncontrollable heart failure, angina, hypertension, arrhythmia
9. With severe neurological/psychological symptoms
10. With watery diarrhea
11. Pregnant or lactating women or women with unknown or suspected pregnancy
12. Inappropriate patients for entry on this study in the judgement of the investigator
13. Diagnosed as Resectable/Unresectable pancreatic carcinoma on NCCN guideline (Version 2.2016)

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival time from the first day of protocol therapy | Up to 60 months

SECONDARY OUTCOMES:
Recurrence free survival from the first day of protocol therapy | Up to 60 months
Adverse effect | Up to 30 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
Morbidity based on Clavien Dindo classification of more than Grade3 | Up to 30 weeks
Response rate | Up to 12 weeks
Chemotherapeutic effect grade based on Evans classification | Up to 12 weeks
Resection rate | Up to 30 weeks
R0 resection rate | Up to 30 weeks
Intraoperative blood loss | Up to 30 weeks
The overall morbidity rates based on Clavien Dindo classification | Up to 50 weeks
Number of patient rate in postoperative adjuvant therapy | Up to 30 weeks
Dose intensity | Up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (18):
- Japan (18):
  - Hirosaki University, Hirosaki, Aomori
  - Kobe University, Kobe, Hyōgo
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Nara Medical University, Kashihara, Nara
  - Kansai Medical University, Hirakata, Osaka
  - Kinki University, Sayama, Osaka
  - Osaka University, Suita, Osaka
  - Osaka Medical University, Takatsuki, Osaka
  - Shiga Medical University, Ōtsu, Shiga
  - Chiba University, Chiba
  - Gifu University, Gifu
  - Hiroshima University, Hiroshima
  - Kumamoto University, Kumamoto
  - Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto University, Kyoto
  - Nagoya University, Nagoya, Aichi
  - Osaka City University, Osaka
  - Second Department of Surgery, Wakayama Medical University, School of Medicine, 811-1 Kimiidera, Wakayama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okada KI, Kimura K, Yamashita YI, Shibuya K, Matsumoto I, Satoi S, Yoshida K, Kodera Y, Akahori T, Hirono S, Eguchi H, Asakuma M, Tani M, Hatano E, Ikoma H, Ohira G, Hayashi H, Wan K, Shimokawa T, Kawai M, Yamaue H; NAC-GA investigators. Efficacy and safety of neoadjuvant nab-paclitaxel plus gemcitabine therapy in patients with borderline resectable pancreatic cancer: A multicenter single-arm phase II study (NAC-GA trial). Ann Gastroenterol Surg. 2023 Jul 8;7(6):997-1008. doi: 10.1002/ags3.12712. eCollection 2023 Nov. PMID 37927936